CLINICAL TRIAL: NCT02111434
Title: Phase 4 Study of Effect of Testosteron Treatment on the Visceral Adiposity Index and Triglyceride/High-density Lipoprotein Cholesterol Ratio in the Congenital Hypogonadotropic Hypogonadism
Brief Title: Visceral Adiposity Index and Triglyceride/High-density Lipoprotein Cholesterol Ratio in the Congenital Hypogonadotropic Hypogonadism and Effect of Testosteron Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, cem haymana, MD, Gulhane School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GSM-022014
Record Dates: First submitted 2014-04-05; First posted 2014-04-11 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Hypogonadism
Keywords: visceral adiposity index; triglycerides / hdl cholesterol ratio; testosterone
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- testosterone (Experimental): testosterone gel per day for 6 months testosterone 250 mg injection per 3-4 weeks for 6 months
  Interventions: Drug: Testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone 250 mg injection per 3-4 weeks for 6 months
  Other Names: sustanon 250 mg

SUMMARY:
The study is designed to answer the following questions:

1. What is the levels of visceral adiposity index and Triglycerides/HDL cholesterol ratio in hypogonadism?
2. What is the effect of testosterone replacement on the visceral adiposity index and Triglycerides/HDL cholesterol ratio?

DETAILED DESCRIPTION:
This is a retrospective design, which is performed by investigating the registrations of patients with hypogonadotrophic hypogonadism between the years 2007-2010.

ELIGIBILITY:
Inclusion Criteria:

* Men
* Congenital hypogonadism
* Treatment Naive

Exclusion Criteria:

* Previous history of androgen replacement
* Hypertension
* Diabetes mellitus

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2013-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
time to change of visceral adiposity index with testosteron replacement | baseline and 6 months
time to change of TG/HDL cholesterol ratio with testosteron replacement | baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Gulhane School of Medicine, Ankara, Turkey (Türkiye)